CLINICAL TRIAL: NCT02393898
Title: BELOVA: A Non-Interventional Study to Collect Data on the Safety and Efficacy of Frontline Bevacizumab Treatment in Ovarian Cancer Patients 70 Years and Older
Brief Title: BELOVA Data Collection: Safety and Efficacy of Frontline Bevacizumab Treatment in Participants With Ovarian Cancer 70 Years and Older
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29515
Record Dates: First submitted 2015-03-12; First posted 2015-03-20 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Elderly Participants with Ovarian Cancer: Elderly participants aged 70 years and older administered frontline treatment for International Federation for Gynecology and Obstetrics (FIGO) stage IV epithelial ovarian, fallopian tube, or primary peritoneal cancer with bevacizumab in combination with chemotherapy according to standard of care.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be prescribed by the local clinician according to the SmPC and standard of care for up to 15 months. No treatment will be provided by the Sponsor in this non-interventional study.
  Other Names: Avastin
Drug: Carboplatin — Carboplatin will be prescribed by the local clinician according to local labeling and standard of care for up to 18 weeks. No treatment will be provided by the Sponsor in this non-interventional study.
Drug: Paclitaxel — Paclitaxel will be prescribed by the local clinician according to local labeling and standard of care for up to 18 weeks. No treatment will be provided by the Sponsor in this non-interventional study.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy in the frontline treatment of ovarian cancer in participants 70 years of age and older in routine clinical practice in Belgium. Bevacizumab will be used in combination with carboplatin/paclitaxel followed by bevacizumab as maintenance in accordance with the Summary of Product Characteristics (SmPC).

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years and older
* No treatment with any other investigational agent within 28 days or 2 half-lives (whichever is longer) prior to enrollment

Exclusion Criteria:

* Contraindications, warnings, and precautions for bevacizumab

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Real-world patients (70 years of age and older) with epithelial ovarian, fallopian tube, or primary peritoneal cancer who are receiving frontline treatment with bevacizumab and chemotherapy according to standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Per routine clinical practice during bevacizumab treatment (up to 15 months)
Time to First Incidence of Adverse Events of Special Interest | Per routine clinical practice during bevacizumab treatment (up to 15 months)

SECONDARY OUTCOMES:
Progression-Free Survival According to Response Evaluation Criteria in Solid Tumors (RECIST) | Per routine clinical practice during bevacizumab treatment (up to 15 months) and at 6 and 12 months after end of bevacizumab (approximately 27 months overall)
Percentage of Participants with Complete or Partial Response According to RECIST | Per routine clinical practice during bevacizumab treatment (up to 15 months) and at 6 and 12 months after end of bevacizumab (approximately 27 months overall)
Overall Survival | Per routine clinical practice during bevacizumab treatment (up to 15 months) and at 6 and 12 months after end of bevacizumab (approximately 27 months overall)
Comprehensive Geriatric Assessment Subscale Scores | Baseline, end of chemotherapy (up to 18 weeks), and after 10 and 15 months of bevacizumab treatment or at disease progression (up to 15 months overall)
Dosage of Bevacizumab in Milligrams per Kilogram (mg/kg) | Every 3 weeks according to SmPC for up to 15 months
Total Number of Bevacizumab Doses | Every 3 weeks according to SmPC for up to 15 months
Percentage of Participants by Chemotherapy Used in Combination with Bevacizumab | Every 3 weeks per routine clinical practice for up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Belgium (26):
  - Onze Lieve Vrouwziekenhuis Aalst, Aalst
  - AZ Sint Lucas Brugge, Assebroek
  - Imeldaziekenhuis, Bonheiden
  - AZ KLINA, Brasschaat
  - AZ Sint Jan, Bruges
  - CHU St Pierre (St Pierre), Brussels
  - Cliniques Uni Ires Saint-Luc; Gynaecology, Brussels
  - GHdC Site Notre Dame, Charleroi
  - UZ Antwerpen, Edegem
  - ZOL (Sint Jan), Genk
  - AZ Maria Middelares, Ghent
  - AZ Sint Lucas (Sint Lucas), Ghent
  - UZ Gent, Ghent
  - CH Jolimont - Lobbes (Jolimont), Haine-Saint-Paul
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
  - Chr de La Citadelle, Liège
  - CHU Sart-Tilman, Liège
  - Clinique Saint-Joseph, Liège
  - Clinique Ste-Elisabeth, Namur
  - AZ Damiaan, Ostend
  - AZ Nikolaas (Sint Niklaas), Sint-Niklaas
  - AZ Turnhout Sint Elisabeth, Turnhout
  - CHR de Verviers - East Belgium, Verviers
  - Sint Augustinus Wilrijk, Wilrijk

REFERENCES:
- [Derived] Vergote I, Van Nieuwenhuysen E, De Waele S, Vulsteke C, Lamot C, Van den Bulck H, Claes N, Graas MP, Debrock G, Spoormans I, Vuylsteke P, Honhon B, Verhoeven D, De Maeseneer D, Dirix L, Mebis J, Vroman P, Denys H, Martinez Mena C, Pelgrims G, Van Steenberghe M, van Gorp T, Gennigens C. Prospective non-interventional BELOVA/BGOG-ov16 study on safety of frontline bevacizumab in elderly patients with FIGO stage IV ovarian cancer: a study of the Belgian and Luxembourg Gynaecological Oncology Group. Int J Gynecol Cancer. 2022 Jun 6;32(6):753-760. doi: 10.1136/ijgc-2021-003190. PMID 35063943